CLINICAL TRIAL: NCT03581006
Title: Food Intake REstriction for Health OUtcome Support and Education (FIREHOUSE) Trial
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-00127
Record Dates: First submitted 2018-06-15; First posted 2018-07-10 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Lung Injury; Particulate Matter Inhalation Injury
Keywords: World Trade Center; Firefighters; FDNY; 9/11; Metabolomics; FIREHOUSE
MeSH Terms: conditions — Lung Injury | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — FEV1<LLN to define WTC-LI; resistant subjects had an FEV1>= LLN at all timepoints post 9/11.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: This observational cohort study will follow firefighters enrolled in Monitoring and Treatment Program. Investigators will include firefighters in the validation cohort who were present at the WTC site within 3 days of 9/11, have consent, and have abnormal post-9/11 lung function.
  This intervention group will undergo technology based monitoring and behavioral participation in a dietary and exercise program with the intent of weight loss and compliance with a low-calorie Mediterranean diet.
  Interventions: Dietary Supplement: Low-Calorie Mediterranean Diet; Combination Product: Technology based monitoring and behavioral participation
- Control (Usual care) Group: This observational cohort study will follow firefighters enrolled in Monitoring and Treatment Program. Investigators will include firefighters in the validation cohort who were present at the WTC site within 3 days of 9/11, have consent, and have abnormal post-9/11 lung function.
  This group will receive no dietary or behavioral intervention. They will continue usual care with their home physicians.
  Interventions: Other: Usual care group

INTERVENTIONS:
Dietary Supplement: Low-Calorie Mediterranean Diet — Participants in the intervention group will receive 6 months of education and behavioral counseling with self-monitoring to help them adopt a Mediterranean-style, calorie-restricted diet, and engage in physical activity
  Other Names: LoCalMed
  Groups: Intervention Group
Combination Product: Technology based monitoring and behavioral participation — Intervention participants will use smart phones to connect to intervention applications, WebEx, MyNetDiary
  Other Names: LoCalMed
  Groups: Intervention Group
Other: Usual care group — Control group, who will receive no dietary or behavioral intervention during the trial
  Other Names: Control group
  Groups: Control (Usual care) Group

SUMMARY:
This is a randomized-controlled unblinded clinical trial to investigate dietary intervention on metabolic biomarker assessment in World Trade Center (WTC) Lung Injury (LI) in firefighters. The purpose of this study is to evaluate biomarkers of metabolic dysregulation that have previously been found to predict WTC-LI in a case cohort study selected from the entire exposed firefighter cohort, and attempt to alter these metabolites using dietary intervention and a technology-supported behavioral modification program. Investigators will measure Pre/Post global metabolic expression in WTC-exposed, symptomatic firefighter serum sampled after 6-month intervention, as well as clinical outcomes of WTC-LI in the study group vs controls.

DETAILED DESCRIPTION:
Investigators propose to measure metabolites on this expanded cohort with serum sampled before and after 6-month intervention with calorie restricted Mediterranean diet to: 1) determine the effects of a technology assisted calorie restricted diet on metabolic risk and lung function; 2) determine differences between usual care and intervention group using genomics and metabolomics that may be targetable markers for further evaluation; 3) quantify the metabolome and evaluate pre/post changes in BMI, FEV1, FeNo, vascular stiffness, and overall quality of life; and 4) explore dietary modification as treatment of WTC-LI. The biomarker profile of the cohort control will be useful for discovering biomarker associations with other disease manifestations such as: bronchial wall thickening on CT, obstruction on FEV1 /FVC ratio, bronchodilator response, methacholine reactivity, and other definitions of loss of FEV 1 . This cohort control will be an asset to future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-90.
2. Born male sex and currently identify as genetic male
3. FDNY rescue and recovery worker.
4. Documented WTC exposure.
5. Enrolled in the FDNY WTC Health Program
6. Subjects are willing and able to consent for themselves to study enrollment
7. Subjects are willing and able to participate in study procedures
8. Are able to perform their activities of daily living independently
9. Are either light duty or retired FDNY Firefighters
10. Have an FEV1 less than the LLN of predicted for age/sex/weight documented at any time after 9/11/2001.
11. Have a BMI>27 kg/m2 and <50kg/m2
12. Willing and able to modify their diet and activity level.
13. Subjects who have a spirometry available within the last 36 months, and at their post-9/11 visits at the FDNY
14. Demonstrate minimal proficiency using a smart phone
15. Have means to accommodate transportation to/from in-person visits

Exclusion Criteria:

1. Have pre-existing and documented conditions or concurrent diagnoses, including (and not necessarily limited to) active cancer, severe heart disease, significant cognitive impairment, eating disorders, significant psychiatric illness, end-stage COPD, severe pulmonary hypertension, or organ transplant.
2. Concomitant use of interfering medication(s) or devices currently or within the month prior to enrollment, including anti-retrovirals, human monoclonal antibodies, supplemental daytime oxygen, and insulin pumps.
3. Severe gastrointestinal issues or illnesses that would prevent adherence to the proposed diets.
4. Severe kidney disease requiring dialysis
5. Severe liver disease requiring frequent medical intervention
6. Participating in other diet modification studies.
7. High dose steroid (>20mg prednisone or equivalent) or other hormonal treatments/chemotherapy use in the last month, including testosterone supplementation.
8. Life-expectancy < 6 months
9. BMI ≥50 kg/m2 or ≤27 kg/m2
10. Recent significant intentional or unintentional weight loss, defined as over 5% reduction in total body weight over the last month. (Blackburn Criteria).
11. Significant or severe alcohol abuse disorder

Ages: 21 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only
Study Population: FDNY rescue and recovery worker with 9/11 exposure with documented WTC-LI by spirometry criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | 4 Years
  Body mass (weight in kg) divided by square of the body height (measured in meters), expressed in units kg/m^2

SECONDARY OUTCOMES:
Pulmonary Function using FEV Measure | 4 Years
  Forced expiratory volume (FEV) using spirometer that measures the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled.
St. George's Respiratory Questionnaire (SGRQ) | 4 Years
  Airways-disease specific paper questionnaire assessing symptoms, effect on activity level, and impact on quality of life.
Electrocardiogram (EKG) | 4 years
  Non-invasive brief electrical recording of heart rate and rhythm using electrodes placed on the chest
Fraction of exhaled nitrous oxide (FENO) | 4 years
  Simple breathing test to measure airway inflammation as often seen in asthma or particulate matter lung injury, measured in ppb.
Pulse Wave Velocity (PWV) | 4 years
  Non-invasive measurement to ascertain vascular stiffness, by measuring the velocity at which the blood pressure pulse propogates through the circulatory system. This is done using a simple non-invasive blood pressure cuff assessment at the carotid and femoral arteries. It is measured as a velocity, in meters/per second.
Individual microbiome profile - stool sample | 4 years
  Simple home collection of a stool sample using a sterile collection kit, provided to the human subject. Stool will be used to generate a microbiome profile unique to that individual, reported as bacterial species found in the gut flora, that may predict lung injury. There is no risk to the human subject aside that of providing a stool sample. All individual information is de-identified for personal protection.
6-minute walk test (6MWT) | 4 years
  Simple exercise capacity assessment measuring distance walked over 6 minutes, measured in meters.
Individual metabolomic profile - blood sample | 4 years
  Routine blood testing via sterile phlebotomy to assess metabolic biomarkers that may or may not predict lung injury. These metabolites are generated in all individuals based on their dietary and exercise habits, underlying comorbidities, and unique metabolism. Measured in routine blood samples, and quantified based on unique chemical composition of that molecule. There is no additional risk to the human subject aside that of venipuncture.
Individual genomic profile - saliva sample | 4 years
  Simple home collection of sputum/saliva sample using a buccal swab kit, provided to the human subject. Saliva will be used to generate a genetic profile unique to that individual, reported as chromosomes, genes, and proteins that may predict lung injury. There is no risk to the human subject aside that of providing a sputum sample. All individual information is de-identified for personal protection.
Short-form-36 (SF-36) questionnaire | 4 years
  Generalized paper questionnaire for self-assessment of mental health, general health perception, and overall quality of life
Routine vital signs - Heart Rate | 4 years
  Brief assessment of heart rate (pulse) measured in beats/per minute
Routine vital signs - Blood Pressure | 4 years
  Subjects who have spirometry available within the last 36 months, and at their post-9/11 visits at the FDNY.
Routine vital signs - Body temperature | 4 years
  Brief assessment of body temperature using a basic thermometer under the tongue, measured in degrees Fahrenheit
Neck circumference | 4 years
  Assessment of neck circumference using basic measuring tape, recorded in centimeters
Waist circumference | 4 years
  Assessment of waist circumference using basic measuring tape, recorded in centimeters
Bioelectrical impedance analysis (BIA) | 4 years
  Assessment of lean body mass and total body fat percentage using an InBody bioelectrical impedance analysis scale.
Food Frequency Questionnaire | 4 years
  Paper assessment of typical dietary intake over previous one month, multiple choice answers

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nolan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States